CLINICAL TRIAL: NCT02631187
Title: Feasibility Study of Balloon Eustachian Tuboplasty (BET) for Grade 2 and 3 Pars Tensa Retractions
Brief Title: Feasibility Study of Balloon Eustachian Tuboplasty (BET)
Acronym: BET
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit any trial partcipants
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15/P/164
Record Dates: First submitted 2015-12-01; First posted 2015-12-16 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2016-10

CONDITIONS: Retraction of the Pars Tensa of the Tympanic Membrane; Eustachian Tube Dysfunction; Retraction Pocket of the Tympanic Membrane
Keywords: Grade 2 retraction of the pars tensa of the tympanic membrane; Grade 3 retraction of the pars tensa of the tympanic membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon Eustachian Tuboplasty (Experimental): Balloon Eustachian tuboplasty = dilatation of the cartilaginous Eustachian tube with a balloon catheter device performed with endoscopic control under general anaesthetic
  Interventions: Device: Bielefeld balloon

INTERVENTIONS:
Device: Bielefeld balloon — Balloon Eustachian tuboplasty = dilatation of the cartilaginous Eustachian tube with a balloon catheter device performed with endoscopic control under general anaesthetic

SUMMARY:
This is a study that aims to evaluate the feasibility of undertaking a United Kingdom (UK) multi-centre randomised controlled trial of BET for the treatment of moderate (grade 2 or 3) retraction pockets (RPs). This future study will aim to address the question: Does BET improve symptoms scores, audiometry and otoscopic appearance of Grade 2-3 pars tensa RPs in adult patients?

Currently conservative treatments for this condition has been shown to be ineffective; there is a significant risk of progression to hearing loss or more serious complications in untreated retraction pockets; and the surgical treatments available to us in the UK not only have a number of risks and drawbacks, but also do not aim to treat the underlying cause (Eustachian Tube dysfunction (ETD)).

ELIGIBILITY:
Inclusion Criteria:

Adult patients over 18 years old with grade 2-3 retraction pocket of the tympanic membrane as assessed by study clinician.

Exclusion Criteria:

* Craniofacial abnormalities (assessed by history and examination)
* Cholesteatoma (assessed by history, otoscopy, tympanogram, PTA)
* Nasopharyngeal tumours (assessed by flexible nasendoscopy)
* Adenoid hypertrophy (assessed by flexible nasendoscopy)
* Patulous ET (assessed by history, otoscopy and tympanogram)
* Previous middle ear surgery (assessed by history and otoscopy)
* Concurrent use of anticoagulant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Acceptability | 6 months
  Acceptability of the procedure, which will be assessed with pre- and post-procedure using the the seven-item Eustachian Tube Dysfunction Questionnaire (ETDQ-7).
Patient Focus Group | 6 months
  Thematic analysis of Patient Focus Group discussions. Standardised questions and focus group discussion with patients with (i) un-operated asymptomatic Retraction Pockets (RPs), (ii) un-operated symptomatic RPs, (iii) RPs treated with cartilage tympanoplasty, and (iv) RPs treated with BET. These will qualitatively assess (as appropriate) positive and negative aspects of patient experience, such as living with the RP, the procedure itself, their recovery, any after effects, and participating in the study. Focus groups will consist of 6 patients in each group.
Complications | 6 months
  An assessment of the number of complications in the 20 participants undergoing BET will also be performed as a marker of safety of the procedure.

SECONDARY OUTCOMES:
Demand | 1 year
  Demand assessed by recruitment rate
Cost analysis of treatment | 1 year
  Cost analysis of BET vs. cartilage tympanoplasty
Comparison of otoendoscopy images | Assessed pre-intervention and post-intervention at 2 weeks and 6 months.
  Comparison of otoendoscopy images by two experienced observers and computer software (ImageJ). Assessed pre-intervention and post-intervention at 2 weeks and 6 months.
Ability to perform Valsalva | Assessed pre-intervention and post-intervention at 2 weeks and 6 months.
  Ability to perform Valsalva measured as always, sometimes or never. Assessed pre-intervention and post-intervention at 2 weeks and 6.
Tympanometry | Assessed pre-intervention and post-intervention at 2 weeks and 6 months.
  Tympanometry (peak middle ear pressure and compliance, and Jerger grade (Improved, unchanged, worse)). Assessed pre-intervention and post-intervention at 2 weeks and 6 months.
pure-tone average (PTA) hearing loss | Assessed pre-intervention and post-intervention at 2 weeks and 6 months.
  PTA (air conduction at 0.25, 0.5, 1, 2, 3, 4, 6, 8kHz; bone conduction at 0.5, 1, 2, 3, 4 kHz) with calculation of air bone gap at 0.5, 1, 2, 3 and 4kHz. Assessed pre-intervention and post-intervention at 2 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James Rainsbury, BMBS MSc FRCS, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607